CLINICAL TRIAL: NCT03048136
Title: A Phase Ib/II Safety Trial of Nivolumab in Combination With Ipilimumab Administered in Participants With Chemotherapy-naive Stage IV or Recurrent Non-small Cell Lung Cancer (NSCLC) (CheckMate 955: CHECKpoint Pathway and nivoluMAb Clinical Trial Evaluation 955)
Brief Title: A Safety Study of Nivolumab in Combination With Ipilimumab in Participants With Advanced Non-small Cell Lung Cancer
Acronym: CheckMate 955
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Business objective has changed
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-955
Record Dates: First submitted 2017-02-08; First posted 2017-02-09 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Flat-Dose (Experimental): Nivolumab flat dose + Ipilimumab
  Interventions: Drug: Nivolumab; Drug: Ipilimumab
- Weight-Based Dose (Experimental): Nivolumab weight-based dose + Ipilimumab
  Interventions: Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Nivolumab — Specified dose on specified days
  Other Names: BMS-936558; Opdivo
Drug: Ipilimumab — Specified dose on specified days
  Other Names: BMS-734016; Yervoy

SUMMARY:
A Study to Evaluate Safety in Participants with Chemotherapy-naïve Stage IV or Recurrent Non-small Cell Lung Cancer Treated With Nivolumab in Combination with Ipilimumab

DETAILED DESCRIPTION:
A Study to Evaluate Safety in Participants with Chemotherapy-naïve Stage IV or Recurrent Non-small Cell Lung Cancer Treated With Nivolumab in Combination with Ipilimumab

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* 1) Stage IV or recurrent non-Small cell lung cancer
* 2) Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1
* 3) Prior adjuvant or neoadjuvant chemotherapy for local, advanced disease allowed if completed at least 6 months prior to randomization

Exclusion Criteria:

* 1) Known epidermal growth factor receptor (EGFR) mutations or anaplastic lymphoma syndrome(ALK) translocations that are sensitive to targeted inhibitor therapy
* 2) Active, known or suspected autoimmune disease or HIV infection
* 3) Prior treatment with any drug that targets T cell co-stimulation pathways (such as checkpoint inhibitors)
* 4) Untreated Central Nervous System metastases

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03-09 (Estimated); Primary Completion 2019-09-29 (Estimated); Study Completion 2019-09-29 (Estimated)

PRIMARY OUTCOMES:
Incidence of high grade (Grade 3-4 and Grade 5) treatment-related select adverse events | Approximately 3 months
Incidence of high grade (Grade 3-4 and Grade 5) immune-mediated adverse events | Approximately 3 months

SECONDARY OUTCOMES:
Progression-free survival (PFS) as determined by the investigator using Response Evaluation Criteria in Solid Tumors (RECIST v1.1) | Up to 24 months
Objective Response Rate (ORR) as assessed by the Investigator using tumor progression per Response Evaluation Criteria in Solid Tumors (RECIST v1.1) | Up to 24 months
Overall survival (OS) as defined as the time from first dosing to the date of death | Up to 5 years
Duration of Response (DOR) as assessed by the investigator using Response Evaluation Criteria in Solid Tumors (RECIST v1.1) | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (16):
- United States (9):
  - Local Institution, San Francisco, California
  - Local Institution, Lincoln, Nebraska
  - Local Institution, Hackensack, New Jersey
  - Local Institution, Columbus, Ohio
  - Local Institution, Lancaster, Pennsylvania
  - Local Institution, Langhorne, Pennsylvania
  - Local Institution, Sayre, Pennsylvania
  - Local Institution, Charleston, South Carolina
  - Local Institution, St. George, Utah
- Local Institution, Viedma, Río Negro Province, Argentina
- Local Institution, Montreal, Quebec, Canada
- Germany (4):
  - Local Institution, Dresden
  - Local Institution, Gauting
  - Local Institution, Gerlingen
  - Local Institution, Großhansdorf
- Local Institution, Lima, Peru

REFERENCES:
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx